CLINICAL TRIAL: NCT04349397
Title: Use of Analgesics and Pain Scores After Pediatric Adenotonsillectomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Christine Martin, Principal Investigator, Oregon Health and Science University
Other Study IDs: 19199
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Pain, Postoperative; Obstructive Sleep Apnea of Child
Keywords: tonsillectomy; adenotonsillectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric tonsillectomy patients: All patients enrolled into study prior to undergoing tonsillectomy or adenotonsillectomy
  Interventions: Behavioral: Medication Tracking Form

INTERVENTIONS:
Behavioral: Medication Tracking Form — Parents will complete medication tracking form for 5 days after child's surgery. They will track medications administered, pain scores, nausea and vomiting

SUMMARY:
The purpose of the study is to quantify the use of pain medications given to children aged 3 - 12 years as well as their pain level through pain scores after they have undergone a tonsillectomy or adenotonsillectomy surgery at Doernbecher Children's Hospital (DCH). We would like to learn more about the pain medications given and the pain scores of children post-surgery for the first 5 days following discharge from the hospital.

DETAILED DESCRIPTION:
You and your child will be enrolled into the study during your child's scheduled surgery at DCH. Your child's surgery, anesthesia plan, and recovery will not change because of your participation in this study. Following discharge from the hospital, the study team will give you two follow-up phone calls that will take approximately 15 minutes. During these phone calls, we will ask you about your child's pain, any nausea or vomiting that has occurred, your child's intake of liquid and food, your child's activity level, and the medications they have been given over the course of the 5 days post-operation. Along with talking over the phone, we will ask you to document this information. After the post-operation day 6 phone call, you and your child will not be asked any additional questions for research purposes and we will ask you to return any documents you were given by the study team. Within 30 days of your and your child's participation in the study, the research team will pull medical information from your child's electronic medical record. Your child's electronic medical record will be reviewed to obtain demographic information such as date of birth, age, weight, ethnicity, medical history, and status information will also be collected such as allergies, potential complications, any pain scores collected during your child's post-anesthesia care unit (PACU) stay, and medical visits. 30 days after your child's surgery, you and your child will no longer be enrolled in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 3-12 that is scheduled to undergo tonsillectomy or adenotonsillectomy, with or without ear tubes or Parent or guardian of a child aged 3-12 years old that is scheduled to undergo tonsillectomy or adenotonsillectomy, with or without ear tubes

Exclusion Criteria:

-

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 1. Parent or guardian refusal of consent
  2. Child has severe OSA (Apnea-Hypopnea Index (AHI) ≥10 or O2 Saturation <85% on polysomnogram)
  3. Child with behavioral disorders (ADHD, ASD, etc.)
  4. Child with genetic disorders (down syndrome, mucopolysaccharidoses, achondroplasia, Prader-Willi syndrome, etc.)
  5. Child with neuromuscular disorders (muscular dystrophy, hypotonia, etc.)
  6. Child with a history of extremely preterm (born at <28 weeks) or very preterm (born at 28-32 weeks)
  7. Child with moderate to severe developmental delay
  8. Child is obese (BMI ≥ 95th percentile)
  9. Child with craniofacial anomalies (retrognathia, micrognathia, midface hypoplasia)
  10. Child with allergies to acetaminophen, ibuprofen, morphine, fentanyl or oxycodone
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Total opioid administered during POD 1-5 (converted to morphine dose equivalents) | POD 1-5
  Total amount of opioid analgesics administered at home on Post-operative days 1-5.

SECONDARY OUTCOMES:
Mean Worst Pain Scores POD 1-5 | POD 1-5
  Average of worst pain scores as documented twice a day on POD 1-5
Total acetaminophen administered on POD 1-5 | POD 1-5
  Total acetaminophen given (total dose and total quantity as mg/kg)
Total ibuprofen administered on POD 1-5 | POD 1-5
  Total ibuprofen given (total dose and total quantity as mg/kg)
Frequency of Vomiting on POD 1-5 | POD 1-5
  Number of days vomiting on POD 1-5
Duration of impaired drinking | POD 1-5
  Return to normal drinking on POD 1-5
Duration of impaired eating | POD 1-5
  Return to normal eating on POD 1-5
Duration of impaired activity | POD 1-5
  Return to normal activity on POD 1-5

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University (OHSU), Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No